CLINICAL TRIAL: NCT02733029
Title: Contrast Enhanced Ultrasonography to Detect Human Renal Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Transplant Nephrologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P000574
Record Dates: First submitted 2016-03-18; First posted 2016-04-11 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Renal Transplant Rejection
MeSH Terms: interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sonazoid contrast (Experimental): The contrast agent Sonazoid will be used during contrast enhanced ultrasonography. This will be a one-time administration of the contrast agent. The contrast agent, Sonazoid (GE Healthcare), is a lipid-stabilized suspension of perfluorobutane microbubbles with a median diameter of 2.4-3.5 μm and will be administered per package insert (intravenously as a continuous infusion). Sonazoid contrast agent will be given at a dose 0.0075 mL/Kg as a bolus intravenous injection while visualizing the kidney transplant.
  Interventions: Drug: Sonazoid; Device: contrast enhanced ultrasonography
- Medical Review (No Intervention): Ultrasound imaging will be taken from a group of subjects recruited for stage 2. These will be obtained through medical record review from subjects with successful renal transplant at BWH and no transplant rejection.

INTERVENTIONS:
Drug: Sonazoid — Sonazoid (GE Healthcare) is a contrast agent that is a lipid-stabilized suspension of perfluorobutane microbubbles
  Arms: Sonazoid contrast
Device: contrast enhanced ultrasonography — Injection of intravenous ultrasound contrast
  Arms: Sonazoid contrast

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of detecting kidney transplant rejection using contrast enhance ultrasonography with the contrast agent Sonazoid.

DETAILED DESCRIPTION:
This study will be divided into two stages. In the first stage the investigators will assess the transplant kidney with ultrasound after contrast injection (Sonazoid) to determine if contrast in the kidney is detectable by ultrasound and to determine if the amount of perfusion can be quantified directly or qualitatively. The investigators aim to have one to two subjects in this stage. If perfusion of the kidney can be assessed, then the investigators will move to stage two of the study.

In stage 2, the investigators will look to determine the ability of the contrast enhanced ultrasonography method to detect renal transplant rejection using Sonazoid. For this stage the investigators will recruit subjects with biopsy confirmed renal transplant rejection. Once subjects are consented, they will undergo contrast enhanced ultrasonography with Sonazoid and have images taken. These images will be compared to images of renal transplant patients that have displayed no rejection or clinical issues. These clinically normal subjects will have previously consented to a medical record review so that the investigators may use their images.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18-75) who have undergone renal transplant at the Brigham and Women's Hospital. [For stage 1 or stage 2]
* Experiencing acute and chronic renal allograft rejection - defined by by examining the histological sections of renal transplant biopsy for a renal pathologist. This is the most accurate way to evaluate the presence of absence of acute and chronic renal transplant biopsy. [For stage 2]
* Adults (ages 18-75) who have undergone renal transplant at the Brigham and Women's Hospital with normal serum creatinine values (~1 mg/dl) [For stage 2 medical record review only]

Exclusion Criteria:

* Hemodynamic instability (e.g., blood pressure < 90)
* Atrial fibrillation with rapid ventricular response
* Arrhythmia
* Poor acoustic windows
* Inability to provide informed consent
* Known right to left or bidirectional cardiac shunts
* Any contraindication such as the history of allergic reactions
* Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Indication of acute renal allograft rejection that has been confirmed by biopsy | Through completion of study, an average of 2 years

SECONDARY OUTCOMES:
Indication of chronic renal allograft rejection (CAN) that has been confirmed by biopsy | Through completion of study, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Reza Abdi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Jeetley P, Hickman M, Kamp O, Lang RM, Thomas JD, Vannan MA, Vanoverschelde JL, van der Wouw PA, Senior R. Myocardial contrast echocardiography for the detection of coronary artery stenosis: a prospective multicenter study in comparison with single-photon emission computed tomography. J Am Coll Cardiol. 2006 Jan 3;47(1):141-5. doi: 10.1016/j.jacc.2005.08.054. Epub 2005 Dec 15. PMID 16386678
- [Background] Tsuruoka K, Yasuda T, Koitabashi K, Yazawa M, Shimazaki M, Sakurada T, Shirai S, Shibagaki Y, Kimura K, Tsujimoto F. Evaluation of renal microcirculation by contrast-enhanced ultrasound with Sonazoid as a contrast agent. Int Heart J. 2010 May;51(3):176-82. doi: 10.1536/ihj.51.176. PMID 20558907
- [Derived] Siedlecki AM, Benson C, Frates M, Azzi J, Hoffman RJ, Milford E, Weins A, Chandraker A, Mc Donald N, Philip White J, Abdi R. First Report of Perfluorobutane Microsphere-Enhanced Ultrasound in the Transplant Kidney. Transplantation. 2019 Oct;103(10):e283-e284. doi: 10.1097/TP.0000000000002856. No abstract available. PMID 31335773